CLINICAL TRIAL: NCT06445322
Title: Prescreening Study to Identify Potential Participants With ABCA4-related Retinopathy for ACDN-01 Clinical Trials
Brief Title: Prescreening Study to Identify Potential Stargardt Participants for ACDN-01 Clinical Trials
Status: Recruiting | Type: Observational
Sponsor: Ascidian Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ACDN-01-000
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stargardt Disease; Stargardt Disease 1; Cone Rod Dystrophy; Juvenile Macular Degeneration
Keywords: ABCA4; ABCA4-related retinopathy; Stargardt Disease; Stargardt macular dystrophy; Cone rod dystrophy; Gene editing; RNA; Gene Therapy; Exon editing; IRD; Inherited retinal disease; Inherited retinal dystrophy; Inherited retinal degeneration
MeSH Terms: conditions — Stargardt Disease; Cone-Rod Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prescreening Group: The prescreening study consists of genetic and visual assessments and will require at least 1 onsite visit. All clinical assessments performed are for the purpose of determining research eligibility for ACDN-01 clinical trials.
  Interventions: Diagnostic Test: Prescreening Assessments

INTERVENTIONS:
Diagnostic Test: Prescreening Assessments — Various genetic and visual assessments.

SUMMARY:
This is an observational prescreening study. Individuals who are eligible for prescreening will undergo testing procedures that may be used to determine eligibility in ACDN-01 clinical trials.

DETAILED DESCRIPTION:
The prescreening process will be used to help determine the initial eligibility and interest of potential participants in ACDN-01 clinical trials by conducting assessments of key eligibility criteria before the clinical trial screening procedures are performed.

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of mutations in the ABCA4 gene
* ABCA4 retinopathy phenotype (Stargardt disease type 1 or cone-rod dystrophy)

Key Exclusion Criteria:

* The presence of pathogenic or likely pathogenic mutations in other genes known to cause cone-rod dystrophy or Stargardt maculopathy
* Retinal disease other than ABCA4-related retinopathy
* Presence of a medical condition (systemic or ophthalmic), psychiatric condition, including substance abuse disorder, or physical examination or laboratory finding that may in the opinion of the principal investigator and sponsor preclude adherence to the scheduled study visits, safe participation in the study, or affect the results of the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females with a diagnosis of ABCA4-related retinopathy will be invited to give informed consent prior to prescreening procedures. After appropriate informed consent/assent has been obtained, potential participants will then undergo the assessments to determine eligibility for ACDN-01 clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Confirm mutations in the ABCA4 gene | 12 months
  Using a Clinical Laboratory Improved Amendments (CLIA)-certified laboratory.
Confirm the absence of pathogenic mutations in genes known to cause retinal disease other than ABCA4-related retinopathy | 12 months
  Using a Clinical Laboratory Improved Amendments (CLIA)-certified laboratory.
Measure BCVA and LLVA | 12 months
  Measure best corrected visual acuity and low luminance visual acuity
Measure the area of retinal atrophy | 12 months
  Using FAF imaging
Measure baseline retinal structure | 12 months
  Using OCT (SD-OCT)
Historical FAF or OCT images | 4 years
  Confirm historical timepoint images
Historical BCVA/LLVA measurements | 4 years
  Collect past measurements

CONTACTS AND LOCATIONS:
Overall Officials: Alia Rashid, Study Director — Ascidian Therapeutics
Locations (8):
- United States (8):
  - University of San Francisco, San Francisco, California
  - Vitreo Retinal Associates, Gainesville, Florida
  - Wilmer Eye Institute at John Hopkins, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Foundation of Texas, Dallas, Texas
  - Retina Consultants of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No